CLINICAL TRIAL: NCT02547896
Title: Effectiveness of Non-steroidal Anti-inflammatory Diclofenac and Its Association to the Opioid Codeine for Pain, Swelling and Trismus in the Bilateral Mandibular Third Molar Extraction With a High Degree of Difficulty Model.
Brief Title: Effectiveness of Diclofenac and Its Association to Codeine After Lower Third Molar Extraction.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Paulo Zupelari Goncalves, DDS., University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 30880914.1.0000.5417
Record Dates: First submitted 2015-09-10; First posted 2015-09-11 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Impacted Third Molar Tooth
Keywords: codeine; diclofenac; impacted third molar tooth
MeSH Terms: interventions — Codeine; Diclofenac; Analgesia; Analgesics, Opioid; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pain control using codeine + diclofenac (Experimental): Fifty healthy volunteers underwent removal of symmetrically positioned lower third molars, receiving for pain relief after the procedure 50mg of codeine + 50mg of diclofenac
  Interventions: Drug: Codeine + Diclofenac
- Pain control using diclofenac (Experimental): Fifty healthy volunteers underwent removal of symmetrically positioned lower third molars, receiving for pain relief after the procedure 50mg of diclofenac
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Codeine + Diclofenac — The patients will receive codeine and diclofenac as pain relief medicine after the surgery
  Other Names: Lower third molar surgery; Pain control; NSAID associated with Opioids
  Arms: Pain control using codeine + diclofenac
Drug: Diclofenac — The patients will receive only diclofenac
  Other Names: Lower third molar surgery; Pain control; NSAID
  Arms: Pain control using diclofenac

SUMMARY:
It will be evaluated the clinical efficacy of Diclofenac 50mg (NSAID) compared to its association with Codeine 50mg (opioid) administered in 50 patients requiring extraction of two third molars. After assessing the research parameters, a comparative data analysis, along with the proper application of statistical tests, will provide the basis for an evaluation of both efficiency medications used.

DETAILED DESCRIPTION:
This research will evaluate the clinical efficacy of Diclofenac 50mg (NSAID) compared to its association with Codeine 50mg (opioid) administered in 50 patients aged less than 18 and requiring extraction of two third molars (with very similar positions, whose degree of difficulty is high). It will be assessed the following parameters: 1) onset and duration of surgery after administration of local anesthetic, 2) open mouth prior to surgery, on the 2nd day after the operation and on the 7th day after surgery (removal points), 3) subjective assessment of pain using a visual analog scale, 4) measurement of facial edema in the second day after the operation and on the 7th day after surgery (as compared with the measurements obtained before surgery) and 5) the incidence, type and severity of adverse reactions. The analysis comparative data, along with the proper application of statistical tests, provide the basis for an evaluation of both efficiency medications used.

ELIGIBILITY:
Inclusion Criteria:

* Impacted lower third molar
* not in use of NSAID or opioids in the last one month

Exclusion Criteria:

* Local anesthetics allergy,
* History of gastrointestinal bleeding or ulcers,
* Kidney disease,
* Asthma,
* Allergy or sensitivity to aspirin or any other NSAID or opioids,
* Pregnant or nursing woman,
* Patients using antidepressant, diuretic or aspirin,
* Patients under treatment to quit drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Higher pain control after lower third molar surgeries with codeine + diclofenac | Seven days after surgery
  Reducing pain is measured by visual analogue scale. It is expected that the visual analogue scale (100 mm) presents lower values in patients that underwent surgeries and received the association of codeine + diclofenac compared to whose received only diclofenac. Evaluated periods were 0, 15, 30, 45 min, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72 and 96 hours.

SECONDARY OUTCOMES:
Adverse effects | Seven days after surgery
  Increased reporting of adverse effects during the postoperative period in patients that received codeine + diclofenac assessed by the information contained in the medical records of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Z Goncalves, DDS, Study Chair — Bauru School of Dentistry - University of Sao Paulo - USP